CLINICAL TRIAL: NCT03451461
Title: Asynchronies During Mechanical Ventilation: Factors Related
Brief Title: Asynchronies During Mechanical Ventilation
Status: Completed | Type: Observational
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Candelaria de Haro, Medical Doctor, Corporacion Parc Tauli
Other Study IDs: Asynchronies
Record Dates: First submitted 2018-02-01; First posted 2018-03-01 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Mechanical Ventilation Complication
Keywords: Asynchronies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — Observational study. Clinical data recorded

SUMMARY:
Invasive mechanical ventilation (IMV) is a life support treatment for patients with acute respiratory failure. The IMV can generate adverse effects that may cause alterations in other organs besides the lung, creating an important problem during ICU stay, hospital stay and years after discharge. These consequences on morbidity and mortality have significant economic and social weight. In the United States the IMV represents 2.7 episodes per 1000 habitants, with an estimated cost of $27,000 million, representing 12% of all hospital expenses. The overall mortality in patients with IMV is 30-35%, increasing with age. Therefore, patients receiving IMV are a high-risk population and with higher costs.

A poor interaction between patient and ventilator during IMV can develop asynchronies. The asynchronies may present in 25% of patients. The majority of studies in ICU patients are limited to a evaluation of short periods of time. Asynchronies identification needs the application of respiratory physiology knowledge and the interpretation of respiratory signals from the ventilator waves. This allows identifying in an easy way different situations of "fight", but it also difficult the identification of situation where asynchronies are less obvious, doing that them remain underdiagnosed. Moreover, asynchronies can be only evaluated during a brief period of time, and it's difficult to know their incidence during all the IMV period and to make adjustments to improve them.

In our centre, it has been developed a continuous monitoring system during IMV which integrates, in real-time, all the information derived from digital monitors and ventilators. It allows a continuous and automatic detection of different events (through an intelligent alarm system) and quantification of asynchronies. It was demonstrated that asynchronies are frequent, that it can be present from the beginning of IMV, that it increase in severe patients under deep sedation and it can increase ICU and hospital mortality.

The investigators can study different factors that can influence over asynchronies development or can improve them.

DETAILED DESCRIPTION:
The aim of this study is to analyze the real incidence of asynchronies of patients undergoing mechanical ventilation and to analyze what factors may have an association with their appearance.

This factors includes factors related with the pulmonary mechanics of each patient and other factors such as the treatment administered, especially drugs with sedative and analgesic effect will be taken into account.

This can help to implement strategies for the improvement of asynchronies.

ELIGIBILITY:
Inclusion Criteria:

* Mechanical ventilation more than 48 hours.
* Included during the first 24 hours of mechanical ventilation.

Exclusion Criteria:

* Less than 18 years old
* Pregnant patients
* Do-not-resuscitate orders
* Admitted for organ donation
* Chest tubes with suspected bronchopleural fistula.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the ICU under mechanical ventilation and monitorized with the Better Care System.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Incidence of asynchronies during mechanical ventilation | during all period of mechanical ventilation up to the study end, approximately december 2018
  Data will be collected through the middleware Better Care, an automatic system of asynchronies detection

SECONDARY OUTCOMES:
Influence of sedation and analgesia in the incidence of asynchronies | during all period of mechanical ventilation up to the study end, approximately december 2018
  percentage of asynchronies (double cycling, ineffective efforts, short cycling, prolonged cycling, asynchrony index), dose in miligrams per kilogram daily of medication and type of medication administered daily.
  Medication data will be collected from the mediacal records daily.
Influence of respiratory mechanics in the incidence of asynchronies | during all period of mechanical ventilation up to the study end, approximately december 2018
  percentage of asynchronies (doublé cycling, ineffective efforts, short cycling, prolonged cycling, asynchrony index, peak pressure in cmH2O, plateau pressure in cmH2O, flow liters/minute, peep in cmH2O, tidal volumen in mililiters, compliance in mililiters/cmH2O, resistances cmH2O/liters per second Respiratory emchanics data will be collected through the middleware Better Care

CONTACTS AND LOCATIONS:
Overall Officials: Lluis Blanch, PhD, Study Director — Director of Institut Parc Tauli
Locations (4):
- Spain (4):
  - Candelaria de Haro, Sabadell, Barcelona
  - Hospital Virgen de las Nieves, Granada
  - Fundació Althaia, Manresa
  - Hospital Universitario Central de Asturias, Oviedo

REFERENCES:
- [Derived] Magrans R, Ferreira F, Sarlabous L, Lopez-Aguilar J, Goma G, Fernandez-Gonzalo S, Navarra-Ventura G, Fernandez R, Montanya J, Kacmarek R, Rue M, Forne C, Blanch L, de Haro C, Aquino-Esperanza J; ASYNICU group. The Effect of Clusters of Double Triggering and Ineffective Efforts in Critically Ill Patients. Crit Care Med. 2022 Jul 1;50(7):e619-e629. doi: 10.1097/CCM.0000000000005471. Epub 2022 Feb 7. PMID 35120043
- [Derived] de Haro C, Magrans R, Lopez-Aguilar J, Montanya J, Lena E, Subira C, Fernandez-Gonzalo S, Goma G, Fernandez R, Albaiceta GM, Skrobik Y, Lucangelo U, Murias G, Ochagavia A, Kacmarek RM, Rue M, Blanch L; Asynchronies in the Intensive Care Unit (ASYNICU) Group. Effects of sedatives and opioids on trigger and cycling asynchronies throughout mechanical ventilation: an observational study in a large dataset from critically ill patients. Crit Care. 2019 Jul 5;23(1):245. doi: 10.1186/s13054-019-2531-5. PMID 31277722